CLINICAL TRIAL: NCT04030923
Title: The Effect of High Frequency Repetitive Transcranial Magnetic Stimulation on Depression in Parkinson's Disease
Brief Title: The Effect of Repetitive Transcranial Magnetic Stimulation (rTMS) on Depression in Parkinson's Disease (PD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Hasan, asmaa mohamed mohamed mahmoud hasan assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: rTMS and depression in PD
Record Dates: First submitted 2019-07-21; First posted 2019-07-24 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Depression in Parkinson's Disease
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real rTMS (Active Comparator): Real rTMS high frequency stimulation (25 HZ), with intensity of 80% of resting motor threshold detected from the hand motor area, with total 2000 pulses on the left DLPFC for 10 consecutive sessions totally over period of 10 days.
  Interventions: Device: repetitive transcranial magnetic stimulation
- sham rTMS (Sham Comparator): Sham rTMS high frequency stimulation (25 HZ), with intensity of 80% of resting motor threshold detected from the hand motor area, with total 2000 pulses with coil perpendicular on scalp over the occipital cortex for 10 consecutive sessions totally over period of 10 days.
  Interventions: Device: repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — By defining intensity of 80% of the resting Motor Threshold detected from motor area for Rt Abductor Pollicis Brevis (APB), we will apply repetitive Transcranial Magnetic Stimulation (rTMS) using 70-mm diameter air-cooled figure-of-8 coil and SuperRapid2 Magnetic Stimulator with high frequency (25Hz), Stimuli will be delivered for total 2000 pulse (divided on 50 trains with 40 pulses per train with inter-train interval 30 seconds) for the left DLPFC (coil placed tangential over the optimal position of 7 cm anterior to hand motor hotspot area detected for Real group and the same coil placed perpendicular with hand of coil pointing upward over occipital cortex for Sham group). Sessions will be consecutive for ten days period with repetition of consecutive 5 sessions as boosting doses on 5 days period over the follow up visits every month for the next 3 months.

SUMMARY:
This study aims to assess the therapeutic role of rTMS on parkinson's patients with depression. Patients diagnosed with Parkinson's Disease and depression will be recruited. All patients will be admitted and will be allocated randomly into two groups one of which will receive real sessions of high frequency rTMS for left dorsolateral prefrontal cortex (DLPFC) for 10 consecutive sessions totally over period of 10 days with repeated booster sessions every month during the period of follow up. The other will receive sham sessions.

DETAILED DESCRIPTION:
This study aims to assess the therapeutic role of rTMS on parkinson's patients with depression. Thirty PD patients with depression using United Kingdom (UK ) bank criteria for PD will be recruited from outpatient clinic in Assiut University. All patients will be admitted at Neuropsychiatric Department, Assiut University Hospital/ Assiut, Egypt.Each patient fulfilled the inclusion criteria as having score more than or equal 14 on Beck Depression Inventory (BDI) will be recruited. The patients will be allocated randomly into two groups one of which will receive real sessions of high frequency rTMS (25 HZ), with intensity of 80% of resting motor threshold detected from the hand motor area, with total 2000 pulses for left DLPFC for 10 consecutive sessions totally over period of 10 days with repeated booster session every month during the period of follow up among three months. The other will receive sham sessions. All subjects will be followed up by selected clinical rating scales at different intervals pre session, post 10 sessions, and after one, two and three months.

ELIGIBILITY:
Inclusion Criteria:

* All patients with Parkinson's Disease who were diagnosed according to UK bank criteria for PD, Aged 45-75 years, with criteria for depression (BDI > or = 14), and consent obtained from the patient or his caregiver.

Exclusion Criteria:

* History of repeated head injury
* History of repeated cerebrovascular strokes
* History of defined encephalitis
* Oculogyric crisis, supranuclear gaze palsy
* Family history of more than one relative
* History of drug intake as antipsychotics or 1-methyl-4-phenyl-1,2,3,6-tetrahydropyridine (MPTP) exposure
* Moderate and Severe depression (Hamilton Depression Rating Scale score >16)
* severe dysautonomia
* Cerebellar signs
* Babinski sign
* Strictly unilateral features after 3 years
* Hydrocephalus or intracranial lesion on neuroimaging
* We also excludes patients with intracranial metallic devices or with pacemakers or any other device.
* patients with cognitive impairment (Mini-Mental Status Examination< 24)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
changes in depression severity measurements | three months
  Depression severity changes measured by Hamilton Depression Rating Scale (HAMD)

CONTACTS AND LOCATIONS:
Overall Officials: Eman Khedr, professor, Study Director — Neurology Department, Faculty of Medicine, Assiut University
Locations (1):
- Assuit University, Asyut, Egypt